CLINICAL TRIAL: NCT03476421
Title: Is R1 Vascular Hepatectomy for Hepatocellular Carcinoma Oncologically Adequate?
Brief Title: R1vascular Hepatectomy for HCC Patients
Status: Completed | Type: Observational
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Principal Investigator, Matteo Donadon, Assistant professor of surgery, staff surgeon, Humanitas Clinical and Research Center
Other Study IDs: HCC R1vasc
Record Dates: First submitted 2018-03-15; First posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- R0 hepatectomy: Those HCC patients operated with standard R0 hepatectomy
  Interventions: Procedure: Hepatic resection
- R1par hepatectomy: Those HCC patients operated with R1par hepatectomy
  Interventions: Procedure: Hepatic resection
- R1vasc hepatectomy: Those HCC patients operated with R1vasc hepatectomy
  Interventions: Procedure: Hepatic resection
- R1par+R1vasc hepatectomy: Those HCC patients operated with both R1par and R1vasc hepatectomy
  Interventions: Procedure: Hepatic resection

INTERVENTIONS:
Procedure: Hepatic resection — Surgery of the liver; removal of a part of the liver

SUMMARY:
Since the previous decade, the authors introduced the R1 vascular (R1vasc) resection for the treatment of hepatocellular carcinoma (HCC), and colorectal liver metastases (Torzilli et al. J Am Coll Surg 2005; Viganò et al. Ann Surg Oncol 2016; Torzilli et al. Surgery 2017). However, oncological reliability of tumor exposure in surgery for HCC remains controversial since it has never been validated. The aim of the study is to determine the oncological adequacy of R1vasc hepatectomy in patients with HCC.

DETAILED DESCRIPTION:
A prospective cohort of patients who underwent hepatectomy for HCC between January 2005 and December 2015 is reviewed. The following definitions are adopted: R0 is any resection with at least 1 mm of negative margin; R1vasc is any resection with tumor exposure due to the detachment from major intrahepatic vessel (1st/2nd order glissonean pedicles and hepatic vein at caval confluence); R1-parenchymal (R1par) is any resection with tumor exposure at parenchymal margin.

ELIGIBILITY:
Inclusion Criteria:

* only patients with a primary untreated HCC were included;
* complete follow-up data with available computed tomography (CT) and/or magnetic resonance imaging (MRI) images showing the first recurrence

Exclusion Criteria:

* patients who underwent vascular resection for direct infiltration of the vessel wall
* patients who had radiofrequency ablation in association to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HCC (hepatocellular carcinoma) who underwent hepatectomy.
Sampling Method: Non-Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Rates of local recurrence | From date of surgery until the date of first documented progression or date of death from any cause, which ever came first assessed up to 72 months
  Calculation of the local recurrence (cut-edge tumor re-growth) of R0, R1par, and R1vasc, and R1par+R1vasc hepatectomy.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Torzilli G, Montorsi M, Donadon M, Palmisano A, Del Fabbro D, Gambetti A, Olivari N, Makuuchi M. "Radical but conservative" is the main goal for ultrasonography-guided liver resection: prospective validation of this approach. J Am Coll Surg. 2005 Oct;201(4):517-28. doi: 10.1016/j.jamcollsurg.2005.04.026. PMID 16183489
- [Result] Torzilli G, Donadon M, Palmisano A, Marconi M, Procopio F, Botea F, Del Fabbro D, Cappellani A, Montorsi M. Ultrasound guided liver resection: does this approach limit the need for portal vein embolization? Hepatogastroenterology. 2009 Sep-Oct;56(94-95):1483-90. PMID 19950814
- [Result] Vigano L, Procopio F, Cimino MM, Donadon M, Gatti A, Costa G, Del Fabbro D, Torzilli G. Is Tumor Detachment from Vascular Structures Equivalent to R0 Resection in Surgery for Colorectal Liver Metastases? An Observational Cohort. Ann Surg Oncol. 2016 Apr;23(4):1352-60. doi: 10.1245/s10434-015-5009-y. Epub 2015 Dec 29. PMID 26714946